CLINICAL TRIAL: NCT03475615
Title: A Randomized Study of the Effect of First-line Intraperitoneal Paclitaxel in Combination With SOX Versus SOX Alone in Gastric Cancer Patients With Malignant Ascites
Brief Title: A Study of Intraperitoneal Paclitaxel in Combination With SOX Compared With SOX Alone in Gastric Cancer With Malignant Ascites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-SOXP
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Gastric Cancer; Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Paclitaxel; S 1 (combination); Tegafur; gimeracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOXP (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Paclitaxel; Drug: S-1 (Tegafur, Gimeracil and Oteracil Porassium Capsules)
- SOX (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: S-1 (Tegafur, Gimeracil and Oteracil Porassium Capsules)

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m2, d1, q3w
Drug: Paclitaxel — 40mg/m2 ip，d1、8 ,q3w
  Arms: SOXP
Drug: S-1 (Tegafur, Gimeracil and Oteracil Porassium Capsules) — 40mg/m2 Bid po，d1-14,q3w

SUMMARY:
This study is designed to compare the efficacy of intraperitoneal paclitaxel in combination with SOX, with SOX alone in the first-line treatment of gastric cancer with malignant ascites

ELIGIBILITY:
Inclusion Criteria:

* had a histologically proven adenocarcinoma of the gastroesophageal junction, or stomach that was locally advanced (inoperable) or metastatic
* malignant ascites(over pelvic cavity in CT scan and confirmed by cytology)
* an Eastern Cooperative Oncology Group performance status of 0 to 2
* adequate renal, hepatic, and hematologic function

Exclusion Criteria:

* previous chemotherapy or radiotherapy (unless in the adjuvant setting)
* uncontrolled cardiac disease, or other clinically significant, uncontrolled
* coexisting illness or previous or concurrent cancer
* HER2 positive and willing to use trastuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 10 months
  the internal between the date of enrollment and the date of death or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No